CLINICAL TRIAL: NCT01257815
Title: Ranibizumab Treatment of Diabetic Macular Oedema With Bimonthly Monitoring After a Phase of Initial Treatment. A UK, 18-month, Prospective, Open-label, Multicentre, Single-arm, Phase IIIb Study With 12-month Primary Endpoint, Assessing the Efficacy and Safety of Ranibizumab in Patients With Visual Impairment Due to Diabetic Macular Oedema.
Brief Title: Ranibizumab Treatment of Diabetic Macular Oedema With Bimonthly Monitoring After a Phase of Initial Treatment
Acronym: RELIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DGB14; 2010-022616-39 (EudraCT Number)
Record Dates: First submitted 2010-12-08; First posted 2010-12-10 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Diabetic Retinopathy; Macular Oedema
Keywords: Diabetes mellitus; Diabetic retinopathy; Macular oedema; Visual acuity
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema; Diabetes Mellitus | interventions — Ranibizumab

ARMS (1):
- Ranibizumab 0.5mg (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
This study evaluates a new investigational treatment regimen of three consecutive monthly doses of ranibizumab followed by an as-needed treatment regimen, with monthly follow-up for the first three months then two-monthly follow-up until 18 months in patients with visual impairment due to diabetic macular oedema.The aim of the study is to determine if this treatment regimen is effective and safe in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes mellitus.
* Patients with visual impairment due to focal or diffuse diabetic macular oedema (DMO), and not other causes, in at least one eye who are eligible for laser treatment in the opinion of the investigator.
* Best Corrected Visual Acuity between 78 and 24 letters in the study eye using Early Treatment Diabetic Retinopathy Study (ETDRS)-like grading charts (approximate Snellen equivalent of 20/32 to 20/320).
* Increased central retinal thickness which, in the opinion of the investigator, is due to DMO.

Exclusion Criteria:

* Concomitant conditions in the study eye that could prevent the improvement of visual acuity on study treatment.
* Active intraocular inflammation (grade trace or above) or infection in either eye at enrollment.
* History of uveitis in either eye at any time.
* Structural damage within 0.5 disc diameters of the centre of the macular in the study eye likely to preclude improvement in visual acuity following resolution of macular oedema.
* Planned medical or surgical intervention during the 18-month study period.
* Uncontrolled glaucoma in either eye at screening.
* Blood pressure systolic > 160 mmHg or diastolic > 100 mmHg at screening.
* Ocular conditions in the study eye that require chronic concomitant therapy with topical ocular or systemically administered corticosteroids.
* History of acute thromboembolic event within 4 months of screening.
* Untreated diabetes mellitus.
* Evidence of advanced, severe or unstable concomitant disease or its treatment which may interfere with evaluations or put the patient at special risk.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The change in mean Best Corrected Visual Acuity (BCVA) | Baseline to 12 months

SECONDARY OUTCOMES:
The change in mean Best Corrected Visual Acuity (BCVA) | Baseline to 18 months
Occurrence of ocular and systemic adverse events | Baseline to 18 months
Time course of changes in BCVA | From 6 to 12 and 18 months
Time course of changes in central retinal thickness | From baseline and 6 months to 12 and 18 months
Proportion of patients with 10 and 15 letter improvement or loss in BCVA | From baseline to 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (14):
- United Kingdom (14):
  - Novartis Investigative Site, Torquay, Devon,
  - Novartis Investigative Site, Hull, Hull
  - Novartis Investigative Site, Ayr
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Fife
  - Novartis Investigative Site, Great Yarmouth
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Rugby
  - Novartis Investigative Site, Uxbridge
  - Novartis Investigative Site, York

REFERENCES:
- [Derived] Pearce I, Banerjee S, Burton BJ, Chakravarthy U, Downey L, Gale RP, Gibson J, Pagliarini S, Patel J, Sivaprasad S, Andrews C, Brittain C, Warburton J; RELIGHT Study Group. Ranibizumab 0.5 mg for Diabetic Macular Edema with Bimonthly Monitoring after a Phase of Initial Treatment: 18-Month, Multicenter, Phase IIIB RELIGHT Study. Ophthalmology. 2015 Sep;122(9):1811-9. doi: 10.1016/j.ophtha.2015.05.038. Epub 2015 Jul 3. PMID 26150052